CLINICAL TRIAL: NCT01402765
Title: Interface Pressure Measures for Matresses: a Randomized, Cross-over, Non-inferiority Study Comparing the Nimbus 3 Versus Summit Matresses
Brief Title: Interface Pressure Measures for Matresses: Nimbus 3 Versus Summit
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LOCAL/2011/EV-06; 2011-A00697-34 (Other: ANSM)
Record Dates: First submitted 2011-07-25; First posted 2011-07-26 (Estimated); Last update posted 2025-11-17 (Actual); Status verified 2015-03

CONDITIONS: Chronic Immobile Patients

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Summit first) (Active Comparator): In Group 1 pressure measurements are first taken on the Summit mattress. The patient is then transferred to a Nimbus 3 mattress, and the measures are repeated.
  Interventions: Device: Summit first
- Group 2 (Nimbus 3 first) (Active Comparator): In Group 2 pressure measurements are first taken on the Nimbus 3 mattress. The patient is then transferred to a Summit mattress, and the measures are repeated.
  Interventions: Device: Nimbus 3 first

INTERVENTIONS:
Device: Summit first — Pressure measurements are first taken on the Summit mattress. The patient is then transferred to a Nimbus 3 mattress, and the measures are repeated.
  Arms: Group 1 (Summit first)
Device: Nimbus 3 first — Pressure measurements are first taken on the Nimbus 3 mattress. The patient is then transferred to a Summit mattress, and the measures are repeated.
  Arms: Group 2 (Nimbus 3 first)

SUMMARY:
The primary objective of this study is to compare the distribution of pressure among pressure interfaces between two anti-bedsore mattresses.

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given his/her informed and signed consent
* The patient must be insured or beneficiary of a health insurance plan
* Bedridden patients that still have some measure of mobility, or that can change beds with assistance.
* Patients with symmetrical buttox support
* Body mass index between 16 and 35

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by a previous study
* The patient is under judicial protection, under tutorship or curatorship
* The patient refuses to sign the consent
* It is impossible to correctly inform the patient
* Strict decubitus dorsal position is contra-indicated
* State of agigation or non-cooperation
* Asymetrical deformation of the spine or hips in the frontal plane
* Bed sores present
* Evolving cardiac pathology
* Recent scar at a pressure interface
* Deep vein thrombosis
* Expected life span < 24 weeks

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2012-03; Primary Completion 2012-04-11 (Actual); Study Completion 2012-04-11 (Actual)

PRIMARY OUTCOMES:
Percentage of data capture time at < 30 mmHg (%) | Day 1
  Percentage of data capture time with a pressure redistribution index measured at the sacrum and buttox at < 30 mmHg

SECONDARY OUTCOMES:
Mean interface pressure (mmHg) | Day 1
  Mean interface pressure (mmHg)
Minimum interface pression (mmHg) | Day 1
  Minimum interface pression (mmHg)
Maximum interface pressure (mmHg) | Day 1
  Maximum interface pressure (mmHg)
Percentage of data capture time where the pressures are changing (%) | Day 1
  Percentage of data capture time where the pressures are changing (%)
Matress tolerance: yes/no | Day 1
  Tolerance of mattress: yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Emilie Viollet, MD, Principal Investigator — Centre Hospitalier Universitaire de Nîmes
Locations (1):
- Centre Hospitalier Universitaire de Nîmes, Nîmes, Gard, France

REFERENCES:
- [Result] de Labachelerie C, Viollet E, Alonso S, Nouvel F, Bastide S, Blot M, Fagart W, Gelis A, Dupeyron A. Comparison of interface pressures in two dynamic pressure ulcer prevention supports (NIMBUS 3 and SUMMIT): A randomized controlled trial. J Tissue Viability. 2022 Feb;31(1):11-15. doi: 10.1016/j.jtv.2021.09.002. Epub 2021 Sep 11. PMID 34598852